CLINICAL TRIAL: NCT01571674
Title: Validation of a Clinical Prediction Rule to Identify Patients With Shoulder Pain Likely to Benefit From Cervicothoracic Manipulation: A Randomized Clinical Trial
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Virginia Commonwealth University (Other); University of Colorado, Boulder (Other); Northern Navajo Medical Center (Unknown); Gundersen Lutheran Health System (Other); Waldron's Peak Physical Therapy (Unknown); Temple University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12-0040
Record Dates: First submitted 2012-03-30; First posted 2012-04-05 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Shoulder Pain
Keywords: Cervical; Clinical Prediction Rule; Exercise; Manipulation; Manual therapy; Mobilization; Physical Therapy; Prognosis; Shoulder pain; Thoracic
MeSH Terms: conditions — Shoulder Pain; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Manipulation + Exercise Group (Experimental): The treatment received by the manipulation+exercise group will differ from the exercise group for the first week only (two treatment sessions). During the first two sessions, patients in the manipulation+exercise group will receive cervicothoracic spine manipulations and range of motion (ROM) exercises only. Beginning on the third session these patients will receive the same exercise program as the exercise group.
  Interventions: Procedure: Manipulation + Exercise Group; Procedure: Exercise Group
- Exercise Group (Active Comparator): The exercise group will be treated with a stretching and strengthening program.
  Interventions: Procedure: Exercise Group

INTERVENTIONS:
Procedure: Manipulation + Exercise Group — First 2 sessions
  * High-velocity, low-amplitude manipulations to the thoracic spine.
  * Low-velocity mid to end-range mobilizations to the cervical spine.
  * Active Range of Motion Exercises for the cervicothoracic spine
  Final 6 sessions
  ◦ Evidence based shoulder girdle exercise program
  Arms: Manipulation + Exercise Group
Procedure: Exercise Group — First 2 sessions
  ◦ Active Range of Motion Exercises for the cervicothoracic spine
  Final 6 sessions
  ◦ Evidence based shoulder girdle exercise program

SUMMARY:
The purpose of this study is to determine the validity of previously identified prognostic variables that may identify patients with shoulder pain that are likely to benefit from cervicothoracic spine manipulation.

DETAILED DESCRIPTION:
The investigators have recently identified prognostic variables in a preliminary Clinical Prediction Rule (CPR) that are purported to identify patients with shoulder pain who respond favorably to cervicothoracic spinal manipulative therapy (SMT) and daily home exercises of cervical and thoracic active range of motion exercises. These prognostic variables have been identified in a single study, and therefore it is not known if these factors will be valid in a different group of patients, even ones with similar characteristics as those used in the investigators' initial exploratory study. Further study of these identified factors is needed for validation in an independent sample of patients, which will improve generalizability for clinical practice. In this study, patients with a primary complaint of shoulder pain will be randomly assigned to receive cervicothoracic spine manipulation followed by therapeutic exercises or therapeutic exercise alone. If the variables are in fact meaningful, patients who exhibit 3 or more of the identified prognostic variables and receive cervicothoracic SMT should experience improved outcomes compared to patients who have less than 3 of these variables and receive the same intervention. Additionally, patients who exhibit 3 or more of the identified variables that receive cervicothoracic SMT should also have superior outcomes to patients who exhibit 3 or more of the identified variables and receive an alternate intervention (exercise only). Finally, the investigators will determine if the addition of cervicothoracic SMT to exercise improves outcomes as compared to exercise alone.

ELIGIBILITY:
Inclusion Criteria:

1. Primary complaint of shoulder pain (defined as pain between the neck and the elbow at rest or during movement of the upper arm, see diagram to the right)
2. Age between 18-65 years old
3. Shoulder Pain and Disability (SPADI) score > 20 points

Exclusion Criteria:

1. Medical red flags noted in the patient's Medical Screening Questionnaire (i.e. tumor, fracture, metabolic diseases, RA, osteoporosis, prolonged history of steroid use, etc.)
2. Acute fractures in the shoulder region.
3. Acute severe trauma in the cervical or thoracic region in the last 6 weeks.
4. Contraindications to manipulative therapy (for example osteoporosis of the cervicothoracic spine).
5. Evidence of central nervous system involvement, to include hyperreflexia, sensory disturbances in the hand, intrinsic muscle wasting of the hands, unsteadiness during walking, nystagmus, loss of visual acuity, impaired sensation of the face, altered taste, the presence of pathological reflexes (i.e. positive Hoffman's and/or Babinski reflexes), etc.
6. Diagnosis of cervical spinal stenosis or bilateral upper extremity symptoms
7. Two or more positive neurologic signs consistent with nerve root compression, including any two of the following:

   * Muscle weakness involving a major muscle group of the upper extremity
   * Diminished upper extremity muscle stretch reflex (biceps brachii, brachioradialis, or triceps brachii reflexes)
   * Diminished or absent sensation to pinprick in any upper extremity dermatome
8. Prior surgery to the neck or thoracic spine involving fusion or open reduction internal fixation.
9. Insufficient English language skills to complete all questionnaires
10. Inability to comply with treatment and follow-up schedule

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2012-01; Primary Completion 2014-12 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change in Shoulder Pain and Disability Index (SPADI) Score | 1 week, 4 weeks, 6 months
  The SPADI is a 13 item questionnaire. The pain domain consists of five questions and the disability domain consists of eight. Each question refers to the past week.

SECONDARY OUTCOMES:
Change in the Shortened version of the Disability of the Arm, Shoulder and Hand Index (QuickDASH) | 1 week, 4 weeks and 6 months
  The QuickDASH4 is an eleven-item questionnaire that addresses symptoms and physical function in people with any or multiple disorders involving the upper limb.
Global Rating of Change (GROC) | 1 week, 4 weeks, 6 months
  The GROC asks patients to rate whether their health condition has improved or deteriorated over time to determine the efficacy of a particular treatment. Scores range from -7 (a very great deal worse) to zero (about the same) to +7 (a very great deal better). Intermittent descriptors of worsening or improving are assigned values from -1 to -6 and +1 to +6 respectively.
Change in the Numeric Pain Rating Scale (NPRS) | 1 week, 4 weeks, 6 months
  An 11-point NPRS will be used to measure pain intensity. The scale is anchored on the left with the phrase "No Pain" and on the right with the phrase "Worst Imaginable Pain". Patients rate their current level of pain and their worst and least amount of pain in the last 24 hours. The average of the three ratings or any single rating may be used to represent the patient's level of pain.
Change in the Modified Fear-Avoidance Beliefs Questionnaire (FABQ) | 1 week, 4 weeks, 6 months
  The FABQ is a 16-item questionnaire designed to quantify fear and avoidance beliefs in patients with musculoskeletal disorders. The FABQ has two sub-scales, a 7-item scale to measure fear-avoidance beliefs about work and a 4-item scale to measure fear-avoidance beliefs about physical activity. Each item is scored from 0-6 with possible scores ranging between 0-24 and 0-42 for the physical activity and work subscales, respectively, with higher scores representing increased fear-avoidance beliefs.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Mintken, DPT, Principal Investigator — University of Colorado, Denver
Locations (9):
- United States (9):
  - University of Colorado Denver, Aurora, Colorado
  - Waldron's Peak Physical Therapy, Boulder, Colorado
  - Wardenburg Health Center at the University of Colorado, Boulder, Colorado
  - Franklin Pierce University, Concord, New Hampshire
  - Northern Navajo Medical Center, Shiprock, New Mexico
  - Temple University, Philadelphia, Pennsylvania
  - VCUHS- Virginia Commonwealth University Health System, Richmond, Virginia
  - University of Puget Sound, Tacoma, Washington
  - Gundersen Lutheran, Onalaska, Wisconsin

REFERENCES:
- [Background] Mintken PE, Cleland JA, Whitman JM, George SZ. Psychometric properties of the Fear-Avoidance Beliefs Questionnaire and Tampa Scale of Kinesiophobia in patients with shoulder pain. Arch Phys Med Rehabil. 2010 Jul;91(7):1128-36. doi: 10.1016/j.apmr.2010.04.009. PMID 20599053
- [Background] Mintken PE, Cleland JA, Carpenter KJ, Bieniek ML, Keirns M, Whitman JM. Some factors predict successful short-term outcomes in individuals with shoulder pain receiving cervicothoracic manipulation: a single-arm trial. Phys Ther. 2010 Jan;90(1):26-42. doi: 10.2522/ptj.20090095. Epub 2009 Dec 3. PMID 19959652
- [Background] Mintken PE, DeRosa C, Little T, Smith B; American Academy of Orthopaedic Manual Physical Therapists. AAOMPT clinical guidelines: A model for standardizing manipulation terminology in physical therapy practice. J Orthop Sports Phys Ther. 2008 Mar;38(3):A1-6. doi: 10.2519/jospt.2008.0301. Epub 2008 Feb 29. PMID 18349498
- [Background] Bergman GJ, Winters JC, Groenier KH, Pool JJ, Meyboom-de Jong B, Postema K, van der Heijden GJ. Manipulative therapy in addition to usual medical care for patients with shoulder dysfunction and pain: a randomized, controlled trial. Ann Intern Med. 2004 Sep 21;141(6):432-9. doi: 10.7326/0003-4819-141-6-200409210-00008. PMID 15381516
- [Background] Strunce JB, Walker MJ, Boyles RE, Young BA. The immediate effects of thoracic spine and rib manipulation on subjects with primary complaints of shoulder pain. J Man Manip Ther. 2009;17(4):230-6. doi: 10.1179/106698109791352102. PMID 20140154
- [Background] Boyles RE, Ritland BM, Miracle BM, Barclay DM, Faul MS, Moore JH, Koppenhaver SL, Wainner RS. The short-term effects of thoracic spine thrust manipulation on patients with shoulder impingement syndrome. Man Ther. 2009 Aug;14(4):375-80. doi: 10.1016/j.math.2008.05.005. Epub 2008 Aug 15. PMID 18703377
- [Background] Walser RF, Meserve BB, Boucher TR. The effectiveness of thoracic spine manipulation for the management of musculoskeletal conditions: a systematic review and meta-analysis of randomized clinical trials. J Man Manip Ther. 2009;17(4):237-46. doi: 10.1179/106698109791352085. PMID 20140155
- [Derived] Failla MJ, Mintken PE, McDevitt AW, Michener LA. Trajectory of patient-rated outcomes and association with patient acceptable symptom state in patients with musculoskeletal shoulder pain. J Man Manip Ther. 2023 Aug;31(4):279-286. doi: 10.1080/10669817.2022.2137350. Epub 2022 Oct 27. PMID 36300352
- [Derived] Mintken PE, McDevitt AW, Michener LA, Boyles RE, Beardslee AR, Burns SA, Haberl MD, Hinrichs LA, Cleland JA. Examination of the Validity of a Clinical Prediction Rule to Identify Patients With Shoulder Pain Likely to Benefit From Cervicothoracic Manipulation. J Orthop Sports Phys Ther. 2017 Apr;47(4):252-260. doi: 10.2519/jospt.2017.7100. Epub 2017 Mar 3. PMID 28257617
- [Derived] Mintken PE, McDevitt AW, Cleland JA, Boyles RE, Beardslee AR, Burns SA, Haberl MD, Hinrichs LA, Michener LA. Cervicothoracic Manual Therapy Plus Exercise Therapy Versus Exercise Therapy Alone in the Management of Individuals With Shoulder Pain: A Multicenter Randomized Controlled Trial. J Orthop Sports Phys Ther. 2016 Aug;46(8):617-28. doi: 10.2519/jospt.2016.6319. PMID 27477473